CLINICAL TRIAL: NCT06202794
Title: Effects of Transcutaneous Electrical Nerve Stimulation for the Treatment of Pain and Respiratory Function Following Mastopexy With Augmentation: Study Protocol for a Randomized Controlled Trial
Brief Title: TENS for the Treatment of Pain and Respiratory Function Following Mastopexy With Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Finis Terrae University (Other)
Responsible Party: Principal Investigator, Esteban Fortuny, Physical Therapy, Finis Terrae University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18072023
Record Dates: First submitted 2024-01-01; First posted 2024-01-12 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain; Respiratory Complication
Keywords: TENS; Plastic Surgery; Physical therapy modalities
MeSH Terms: conditions — Pain, Postoperative | interventions — Research Design

STUDY DESIGN:
Intervention Model Description: A two-arm, randomized, sham-controlled trial will be conducted with blinded assessors.
Who Masked: Participant, Care Provider, Investigator
Masking Description: After the website (https://www.randomizer.org) generates a number sequence, blind allocation will be performed using consecutively numbered opaque envelopes. The envelopes will be sealed and stored in a secure cabinet. The main investigator will perform sample randomization and blind assignment. The researcher in charge of administering the treatments will open the envelopes immediately prior to the intervention. The patient, researcher and assessor will have no knowledge about the treatment applied (blinding of assessor and subjects). Only the researcher who administers the intervention (active or sham TENS) will have knowledge of the treatment and will instruct the participant not to provide information on the sensation of electrical stimulus to the assessor measuring pain levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): TENS will be initiated one hour after surgery. A portable device with two channels will be used (Neurodyn Portable TENS, Ibramed, Amparo, São Paulo, Brazil). This device will deliver a biphasic, asymmetrical, balanced current, with a frequency of 100 Hz and pulse duration of 100 μs. Four electrodes (5x5 cm) will be positioned on the left and right sides of the spine according to the indicated instructions. The assessor will increase the intensity to promote a strong tingling sensation, reaching the patient's maximum tolerance level without causing discomfort. Emission will be applied in a single session of one continuous hour and the patients will be informed that the sensation may decrease over time. Every 10 minutes, the assessor will ask the patient if there is habituation to the current and will increase the intensity if necessary. TENS will be administered only once for one hour.
  Interventions: Device: Experimental: Experimental group
- Control group (Sham Comparator): Sham TENS will be performed using equipment identical in appearance to active TENS (Neurodyn Portable TENS, Ibramed, Amparo, São Paulo, Brazil) specifically designed for this study. The device will emit an electrical current gradually increased during the first 30 seconds, followed by a gradual decrease over the subsequent 15 seconds reaching an intensity of 0 mA. The device will remain inactive during the rest of the application, but will have a flashing light, giving the patient the appearance that it is active. The assessor will inform the patient that it is possible to feel the sensation of the current or not depending on individual characteristics. This type of equipment is validated and has been used in other studies to facilitate the blinding of participants. Both systems will be calibrated using a digital oscilloscope (DPO 7000, Tektronix Inc., Beaverton, OR, USA).
  Interventions: Device: Sham Comparator: Control group

INTERVENTIONS:
Device: Experimental: Experimental group — TENS will be initiated one hour after surgery. A portable device with two channels will be used (Neurodyn Portable TENS, Ibramed, Amparo, São Paulo, Brazil). This device will deliver a biphasic, asymmetrical, balanced current, with a frequency of 100 Hz and pulse duration of 100 μs. Four electrodes (5x5 cm) will be positioned on the left and right sides of the spine according to the indicated instructions. The assessor will increase the intensity to promote a strong tingling sensation, reaching the patient's maximum tolerance level without causing discomfort. Emission will be applied in a single session of one continuous hour and the patients will be informed that the sensation may decrease over time. Every 10 minutes, the assessor will ask the patient if there is habituation to the current and will increase the intensity if necessary. TENS will be administered only once for one hour.
  Other Names: TENS Experimental group
  Arms: Experimental group
Device: Sham Comparator: Control group — Sham TENS will be performed using equipment identical in appearance to active TENS (Neurodyn Portable TENS, Ibramed, Amparo, São Paulo, Brazil) specifically designed for this study. The device will emit an electrical current gradually increased during the first 30 seconds, followed by a gradual decrease over the subsequent 15 seconds reaching an intensity of 0 mA. The device will remain inactive during the rest of the application, but will have a flashing light, giving the patient the appearance that it is active. The assessor will inform the patient that it is possible to feel the sensation of the current or not depending on individual characteristics. This type of equipment is validated and has been used in other studies to facilitate the blinding of participants. Both systems will be calibrated using a digital oscilloscope (DPO 7000, Tektronix Inc., Beaverton, OR, USA).
  Other Names: Sham TENS Experimental group
  Arms: Control group

SUMMARY:
Background: Pain after breast plastic surgery affects quality of life. Physical therapy offers effective interventions for this condition, such as transcutaneous electrical nerve stimulation (TENS). Although this resource has been used for more than 20 years, no studies have been published that support its use following this type of surgery. Therefore, the aim of the proposed study is to evaluate the effect of TENS on pain intensity in patients undergoing mastopexy with implants, given the existing evidence on the success of TENS for other conditions.

Methods: A two-arm, randomized, sham-controlled trial will be conducted with blinded assessors. The study will be carried out at the Exercise Physiology and Metabolism Lab of Finis Terrae University. Eligible participants will be women undergoing mastopexy with implants invited by a board-certified plastic surgeon. The participants will be randomly assigned to one of two study groups: Group 1 (surgery + TENS) and Group 2 (surgery + sham TENS). TENS will be administered only one hour after surgery and will remain for one hour. Four assessments will be performed: before treatment (T0), immediately after treatment (T1), one hour (T2) and four hours after TENS (T3). The primary outcome will be pain intensity at rest, pain intensity during movement (standardized movements of both arms: anterior flexion, abduction, and external rotation), and during respiratory function tests. Secondary outcome measures will be maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP), and vital capacity (VC).

Discussion In this study, the effects of TENS on patients with pain following mastopexy with implants will be compared to the effects of a sham TENS intervention. This RCT will offer novel evidence on the potential benefits of TENS in terms of pain intensity at rest as well as during movements and respiratory function tests.

Keywords TENS, Mastopexy, Plastic Surgery, Physical therapy modalities, Clinical trial protocol

DETAILED DESCRIPTION:
OBJECTIVES The aim of the study is to evaluate the effectiveness of transcutaneous stimulation therapy (TENS) on acute pain and respiratory function in patients undergoing mastopexy with implants.

THE PRIMARY OBJECTIVE The primary objective is to assess pain intensity at rest during active arm movements (flexion, rotation, and abduction), and during respiratory muscle strength tests using the numeric pain scale (NRS) after surgery, immediately after the application of the therapy, as well as one and four hours after the intervention.

THE SECONDARY OBJETIVE The secondary objective is to evaluate changes in measures of respiratory muscle function, such as maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP), and vital capacity (VC) as well as the consumption of analgesics for pain after surgery, immediately after the application of the therapy, and one and four hours after the intervention.

TRIAL DESIGN A two-arm, randomized, sham-controlled trial (RCT) will be conducted. The participants and assessor will be blinded to the allocation of the patients to the different groups. This study is reported in accordance with the Consolidated Standards of Trial Reporting (CONSORT). The protocol was developed following the recommendations of Standard Protocol Elements: Recommendations for Interventional Trials (SPIRIT).

The study has received approval from the Human Research Ethics Committee of the Eastern Metropolitan Health Service in Santiago, Chile (approval date: July 31, 2023; process N° 20230731) and will be conducted in accordance with the ethical precepts stipulated in the Declaration of Helsinki.

METHODS: PARTICIPANTS, INTERVENTIONS, AND OUTCOMES STUDY SETTING The study will be conducted at the Physical Therapy Department of Finis Terrae University in the city of Santiago, Chile.

Who will take informed consent? All patients included in the study must validate their participation by signing a statement of informed consent following clarifications of the objectives and procedures given by the assessor.

Intervention description The participants will be divided into two groups: Group 1 (TENS) and Group 2 (sham TENS). Simple randomization will be performed to assign each participant to each group.

Treatment will be performed one hour after surgery and both groups will receive an application of active or sham TENS for one hour. Application will be performed in a single session and four assessments will be performed: immediately after surgery (T0), immediately after TENS (T1) as well as one (T2) and four hours (T3) after intervention with TENS.

Anesthesia protocol The anesthesia-sedation protocol and analgesia scheme will be the same for all participants and under the support of a certified anesthesiologist. All surgeries will be performed under general anesthesia. The anesthetic plan will involve 5 to 10 mg/kg fentanyl combined with the use of propofol for anesthetic induction. Maintenance will be performed with 2 to 3% sevoflurane using an oxygen mixture of over 40%. The control of the maintenance of sevoflurane and the oxygen concentration will involve the use of a gas analyzer. A neuromuscular blocker will be used only for anesthetic induction. Blood pressure control will be maintained with the adjustment of sevoflurane and, when necessary, a vasoactive agent. Mean arterial pressure will be maintained between 50 to 100 mmHg.

Postoperative procedure (analgesia) With the aim of standardizing pain management strategies, all participants will receive the same analgesia scheme at the end of the surgery. This will be based on the use of dipyrone (1 g) administered every 6 hours and ketoprofen (100 mg) every 12 hours, both of which will be administered intravenously. Immediately after surgery, an elastic compression breastplate will be placed to support both breasts and adhesive electrodes will be left positioned for the administration of TENS.

Transcutaneous Electrical Nerve Stimulation (TENS) - Experimental group TENS will be initiated one hour after surgery. A portable device with two channels will be used (Neurodyn Portable TENS, Ibramed, Amparo, São Paulo, Brazil). This device will deliver a biphasic, asymmetrical, balanced current, with a frequency of 100 Hz and pulse duration of 100 μs. Four electrodes (5x5 cm) will be positioned on the left and right sides of the spine according to the indicated instructions. The assessor will increase the intensity to promote a strong tingling sensation, reaching the patient's maximum tolerance level without causing discomfort. Emission will be applied in a single session of one continuous hour and the patients will be informed that the sensation may decrease over time. Every 10 minutes, the assessor will ask the patient if there is habituation to the current and will increase the intensity if necessary. TENS will be administered only once for one hour.

Sham transcutaneous electrical nerve stimulation- Control group Sham TENS will be performed using equipment identical in appearance to active TENS (Neurodyn Portable TENS, Ibramed, Amparo, São Paulo, Brazil) specifically designed for this study. The device will emit an electrical current gradually increased during the first 30 seconds, followed by a gradual decrease over the subsequent 15 seconds reaching an intensity of 0 mA. The device will remain inactive during the rest of the application, but will have a flashing light, giving the patient the appearance that it is active. The assessor will inform the patient that it is possible to feel the sensation of the current or not depending on individual characteristics. This type of equipment is validated and has been used in other studies to facilitate the blinding of participants. Both systems will be calibrated using a digital oscilloscope (DPO 7000, Tektronix Inc., Beaverton, OR, USA).

Both the active and sham TENS treatment groups will have the electrodes positioned in the same place and will undergo all assessments. The researcher who activates the TENS device will not be the same as the one who performs the pain assessments and respiratory function tests. Thus, the assessor will not know which of the study subjects performed treatment with sham or active equipment. The operator who will apply the active and sham TENS treatments will instruct the patient not to give references to the assessor about the sensation of the electrical current.

Sample size The sample size was calculated considering a two-point difference on the NRS between the active TENS and sham groups and a standard deviation of three points based on data from a previous study. For a significance level of 0.05 and 80% statistical power, 37 participants would be needed for each group, constituting a sample n of 74 patients (Minitab, v.15, State College, PA).

The study will include 84 participants (42 per group) in recognition of the crucial role of sample size in determining the power and impact of the study. An additional 15% will be added to the sample size to compensate for possible losses to follow-up (bias due to abandonment). This is consistent with what the literature recommends, which suggests an increase of at least 10% to the sample size, and with the PEDro scale (criterion 8), which advocates for analyzing at least 85% of the data to maintain validity and obtain more robust statistical results and analysis.

Recruitment The participants will be volunteers and will be contacted by the head surgeon, who will initially invite them to participate in the study. The main researcher will contact each of candidate and explain the procedure and objectives of the study. Candidates will then will be asked to sign a statement of informed consent expressing their voluntary desire to participate in the study with the understanding that it is possible to withdraw from the study at any time with no negative consequences.

Assignment of interventions: allocation Sequence generation The patients included will be allocated to one of two groups [Group 1 (active TENS) and Group 2 (sham TENS)] using a simple randomization procedure via the research randomizer website. Block randomization with a 1:1 proportion will be performed, resulting in two groups with equal numbers of women. Each participant will have an equal probability of being randomly allocated to either Group 1 or Group 2.

Concealment mechanism After the website (https://www.randomizer.org) generates a number sequence, blind allocation will be performed using consecutively numbered opaque envelopes. The envelopes will be sealed and stored in a secure cabinet. The main investigator will perform sample randomization and blind assignment. The researcher in charge of administering the treatments will open the envelopes immediately prior to the intervention. The patient, researcher and assessor will have no knowledge about the treatment applied (blinding of assessor and subjects). Only the researcher who administers the intervention (active or sham TENS) will have knowledge of the treatment and will instruct the participant not to provide information on the sensation of electrical stimulus to the assessor measuring pain levels.

Implementation Three independent therapists will work on this study and each will have a specific role. One researcher (R1) will oversee participant recruitment, participant registration, and the random allocation sequence. The interventions will be implemented by a second researcher (R2) (active or sham TENS). All assessments (NRS, MIP, MEP, and VC) will be performed by the main researcher (R3), who will examine and record the data.

Assignment of interventions: blinding Who will be blinded The assessors will be blinded to the assignment of individuals to the different groups and will only be responsible for the assessment procedures. The main researcher responsible for the treatment will not be blinded due to the nature of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* female sex, age between 18 to 55 years in the immediate postoperative period of mastopexy with implants;
* score > 3 for pain intensity on the numeric pain scale (NRS) reported during post-surgery screening;
* no previous experience with the use of TENS or electrical currents for analgesia;
* not having undergone any other type of surgery in the chest region, taking medications to control pain or anxiety, or having a history of pain in the breast region.
* None of the individuals should use bronchodilator therapy or medications that directly act on the respiratory system.

Exclusion Criteria:

* frequent use of bronchodilators, analgesics, muscle relaxants, or psychotropics or allergy to any medication that interferes with surgery (morphine, dipyrone, propofol, lidocaine);
* pregnancy, previous abdominal surgeries, or pre-surgical breast pain;
* any type of inflammatory disease, systemic lupus erythematosus, dermatomyositis or dermatitis in the treatment area, cancer, tumors of any type diagnosed in the previous five years;
* history of epilepsy, metal devices implanted in the body;
* any musculoskeletal injury in the cervical spine, neck or shoulder in the previous three months (fractures, sprains, tendinopathies, dislocations or muscle ruptures) or having a cardiac device, such as an internal automatic defibrillator or pacemaker.
* All patients undergoing combined surgeries or who undergo another surgical procedure in addition to mastopexy with implants or who have knowledge or previous use of TENS or electrical currents for the treatment of pain will be excluded.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at rest | This will be performed at rest immediately after the intervention (T1), 1 hour after treatment (T2) and 4 hour after treatment (T3)
  The primary outcome will be pain intensity, which will be measured using the numeric rating scale (NRS). The NRS is a simple, easy-to-use scale on which the respondent is asked to rate the intensity of current pain using a scale ranging from 0 ("no pain") to 10 ("worst pain imaginable"). This tool has established validity and reliability for measuring acute and postoperative pain intensity. It also has similar sensitivity and correlates to the visual analogue scale.
Pain intensity during movement | This will be performed during movement of arms immediately after the intervention (T1), 1 hour after treatment (T2) and 4 hour after treatment (T3)
  The primary outcome will be pain intensity, which will be measured using the numeric rating scale (NRS). The NRS is a simple, easy-to-use scale on which the respondent is asked to rate the intensity of current pain using a scale ranging from 0 ("no pain") to 10 ("worst pain imaginable"). This tool has established validity and reliability for measuring acute and postoperative pain intensity. It also has similar sensitivity and correlates to the visual analogue scale.

SECONDARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) | Immediately after treatment (T1), 1 h after treatment (T2) and 4 h after treatment (T3)
  To measure inspiratory muscle strength (MIP), the patient will be asked to perform maximal expiration to the residual volume (RV) level and then perform maximal inspiratory effort, which should be maintained for approximately one second.
Maximum Expiratory Pressure (MEP) | Immediately after treatment (T1), 1 h after treatment (T2) and 4 h after treatment (T3)
  To measure expiratory muscle strength (MEP), the patient will be asked to perform maximal inspiration to total lung capacity and then perform maximal expiratory effort, which should be maintained for approximately one second.
Vital Capacity (VC) | Immediately after treatment (T1), 1 h after treatment (T2) and 4 h after treatment (T3)
  Vital capacity (VC) will be measured with the patient in the sitting position using a spirometer (Wright Mark 8) connected to a disposable mouthpiece. A nose clip will be used to prevent air leakage. The test begins with inspiration to total lung capacity, followed by expiration until the residual volume. The highest value of three consecutive measurements will be considered

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Fortuny, PT, Principal Investigator — Finis Terrae University
Locations (1):
- Esteban Fortuny, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Result] da Silva MP, Liebano RE, Rodrigues VA, Abla LE, Ferreira LM. Transcutaneous electrical nerve stimulation for pain relief after liposuction: a randomized controlled trial. Aesthetic Plast Surg. 2015 Apr;39(2):262-9. doi: 10.1007/s00266-015-0451-6. Epub 2015 Feb 10. PMID 25665520
- [Result] DeSantana JM, Santana-Filho VJ, Guerra DR, Sluka KA, Gurgel RQ, da Silva WM Jr. Hypoalgesic effect of the transcutaneous electrical nerve stimulation following inguinal herniorrhaphy: a randomized, controlled trial. J Pain. 2008 Jul;9(7):623-9. doi: 10.1016/j.jpain.2008.01.337. Epub 2008 Apr 3. PMID 18387854
- [Result] Desantana JM, Sluka KA, Lauretti GR. High and low frequency TENS reduce postoperative pain intensity after laparoscopic tubal ligation: a randomized controlled trial. Clin J Pain. 2009 Jan;25(1):12-9. doi: 10.1097/AJP.0b013e31817d1070. PMID 19158541
- [Result] Ducic I, Seiboth LA, Iorio ML. Chronic postoperative breast pain: danger zones for nerve injuries. Plast Reconstr Surg. 2011 Jan;127(1):41-46. doi: 10.1097/PRS.0b013e3181f9587f. PMID 21200198
- [Result] Emmiler M, Solak O, Kocogullari C, Dundar U, Ayva E, Ela Y, Cekirdekci A, Kavuncu V. Control of acute postoperative pain by transcutaneous electrical nerve stimulation after open cardiac operations: a randomized placebo-controlled prospective study. Heart Surg Forum. 2008;11(5):E300-3. doi: 10.1532/HSF98.20081083. PMID 18948245
- [Result] Freynet A, Falcoz PE. Is transcutaneous electrical nerve stimulation effective in relieving postoperative pain after thoracotomy? Interact Cardiovasc Thorac Surg. 2010 Feb;10(2):283-8. doi: 10.1510/icvts.2009.219576. Epub 2009 Nov 12. PMID 19910359
- [Result] Galli TT, Chiavegato LD, Liebano RE. Effects of TENS in living kidney donors submitted to open nephrectomy: a randomized placebo-controlled trial. Eur J Pain. 2015 Jan;19(1):67-76. doi: 10.1002/ejp.521. Epub 2014 May 15. PMID 24831862
- [Result] Galli TT, Chiavegato LD, Santiago NR, Liebano RE. Effects of transcutaneous electrical nerve stimulation on pain, walking function, respiratory muscle strength and vital capacity in kidney donors: a protocol of a randomized controlled trial. BMC Nephrol. 2013 Jan 11;14:7. doi: 10.1186/1471-2369-14-7. PMID 23311705
- [Result] Liebano RE, Vance CG, Rakel BA, Lee JE, Cooper NA, Marchand S, Walsh DM, Sluka KA. Transcutaneous electrical nerve stimulation and conditioned pain modulation influence the perception of pain in humans. Eur J Pain. 2013 Nov;17(10):1539-46. doi: 10.1002/j.1532-2149.2013.00328.x. Epub 2013 May 6. PMID 23650092
- [Result] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Result] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Result] Johnson MI, Paley CA, Jones G, Mulvey MR, Wittkopf PG. Efficacy and safety of transcutaneous electrical nerve stimulation (TENS) for acute and chronic pain in adults: a systematic review and meta-analysis of 381 studies (the meta-TENS study). BMJ Open. 2022 Feb 10;12(2):e051073. doi: 10.1136/bmjopen-2021-051073. PMID 35144946
- [Derived] Pacheco EF, Lyons TV, Liebano RE. Effects of transcutaneous electrical nerve stimulation for the treatment of pain and respiratory function following mastopexy with augmentation: study protocol for a randomized controlled trial. Trials. 2025 Dec 2;27(1):7. doi: 10.1186/s13063-025-09231-9. PMID 41331821

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT06202794/SAP_000.pdf